CLINICAL TRIAL: NCT04784117
Title: Out-of-hospital Cardiac Arrest Epidemiology and Outcomes in Kaunas 2016-2021
Status: Completed | Type: Observational
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Egle Vaitkaitiene (Unknown); Dinas Vaitkaitis (Unknown); Asta Krikscionaitiene (Unknown); Ilona Kajokaite (Unknown); Nerijus Mikelionis (Unknown)
Responsible Party: Principal Investigator, Linas Darginavicius, Principle investigator, Medical director of Emergency department, Lithuanian University of Health Sciences
Other Study IDs: LITOHCA
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subgroup 2016-2018: Subgroup before change of dispatcher protocol
- Subgroup 2019-2021: Subgroup after change of dispatcher protocol
  Interventions: Other: Dispatcher protocol change

INTERVENTIONS:
Other: Dispatcher protocol change — In the beginning of 2019 dispatcher protocol was changed to shorten the time of death detection
  Groups: Subgroup 2019-2021

SUMMARY:
Out-of-hospital cardiac arrest rate is common problem, because of high mortality rate. It is not clear incidence rate, epidemiology and outcomes in Lithuania and Kaunas city included.

DETAILED DESCRIPTION:
This data reported according to UTSTEIN guidelines could be compared with other countries from the region although not much data is available, but it will be a baseline for future references about processes in patient management, demographics, incidence rate and OHCA outcomes.

ELIGIBILITY:
Inclusion Criteria:

* OHCA patients of all ages more than 18 years-old with resuscitation commenced or continued by EMS personnel were included.

Exclusion Criteria:

* obviously dead patients, were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: OHCA patients of all ages more than 18 years-old with resuscitation commenced or continued by EMS personnel
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The detection of death will be shorter | 31 Dec 2021

SECONDARY OUTCOMES:
The survival rate will increase | 31 Dec 2021

CONTACTS AND LOCATIONS:
Locations (2):
- Lithuania (2):
  - Kaunas city ambulance station, Kaunas
  - Lithuanian university of health sciences hospital Kaunas clinics, Kaunas

IPD SHARING:
Plan to Share IPD: Yes
for the purposes of data collection and analysis
Supporting Information: Study Protocol, SAP, CSR, Analytic Code

REFERENCES:
- [Derived] Darginavicius L, Kajokaite I, Mikelionis N, Vencloviene J, Dobozinskas P, Vaitkaitiene E, Vaitkaitis D, Krikscionaitiene A. Short- and long-term survival after out-of-hospital cardiac arrest in Kaunas (Lithuania) from 2016 to 2018. BMC Cardiovasc Disord. 2022 Dec 3;22(1):519. doi: 10.1186/s12872-022-02964-4. PMID 36460967